CLINICAL TRIAL: NCT02317133
Title: Study of the Role of Regulator T Cells in the Pathophysiology of Childhood Henoch Schönlein Purpura
Acronym: FOX-TREG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOIt/2013/TAT-01; 2013-A01264-41 (Other: ANSM)
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2019-03

CONDITIONS: Henoch Schönlein Purpura
Keywords: Tregs; bacterial translocation; cytokines
MeSH Terms: conditions — IgA Vasculitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool samples: DNA extractions for microbiota analysis. Blood samples: DNA extractions for bacterial translocation analysis Blood samples: samples remaining will be kept for further analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HSP: acute episode: Patients in this group are going through an acute episode of Henoch Schönlein Purpura.
  Intervention: Blood samples Intervention: Stool samples
  Interventions: Biological: Blood samples; Biological: Stool samples
- HSP: remission: Patients in this group have had Henoch Schönlein Purpura in the past but currently have no symptoms.
  Intervention: Blood samples Intervention: Stool samples
  Interventions: Biological: Blood samples; Biological: Stool samples
- Control group: Control patients recruited from elective surgery candidates at the participating hospitals.
  Intervention: Blood samples Intervention: Stool samples
  Interventions: Biological: Blood samples; Biological: Stool samples

INTERVENTIONS:
Biological: Blood samples — Compared to routine practice, 3 additional tubes of blood will be drawn for the observational needs of this study.
Biological: Stool samples — Stool samples will be collected for the observational needs of this study (and are not part of routine practice).

SUMMARY:
The primary objective of this study is to search for evidence of quantitative or functional defects in plasma regulatory T cells (Tregs) in pediatric patients with Henoch Schönlein Purpura (HSP) as compared to a control population.

DETAILED DESCRIPTION:
The secondary questions/objectives for this study are:

A. During an inflammatory HSP flare, is there a quantitative and / or qualitative defect in plasma Tregs? Are such blood anomalies real or are they due to a modification of the distribution of theses cells to localized sites? B. In the asymptomatic phase, are there quantitative or functional abnormalities among Tregs in subjects with HSP compared to healthy control subjects? C. Are Treg abnormalities associated with modifications in other blood cell lineages, including B cells secreting IgA and abnormally glycosylated IgA1, and secretion of cytokines during acute relapses and during the asymptomatic phase? D. Can streptococcus or other oral or digestive pathogens (bacterial or viral) (as suggested in other chronic diseases such as rheumatoid arthritis ) provoke (via stimulation Th3) isotype commutation towards secretion of IgA1 at the origin of HSP? Does HSP intestinal damage or imbalance of the intestinal microbiota allow the translocation of intestinal microorganisms that sustain this stimulation?

ELIGIBILITY:
General inclusion criteria for all sub-populations included in the study

* The child (with age- and comprehension-skill-appropriate information) and parents (or persons exercising parental authority) have been informed about the implementation of the study, its objectives, constraints and patient rights
* The child (depending on age) and parents (or persons exercising parental authority) have given their free and informed consent and signed the consent
* The patient must be insured or beneficiary of a health insurance plan

Inclusion criteria for population A: Henoch Schönlein purpura, acute episodes

* The diagnosis of Henoch Schönlein purpura was made by a physician according to the EULAR / PRES / PRINTO 2010 criteria (purpura predominantly on the lower limbs associated with one of the following criteria: abdominal pain, arthralgia or arthritis, kidney damage or suggestive histology (immune deposits dominated by Immunoglobulin A (IgA))
* The patient is not treated via immunosuppression (steroids or other immunosuppressive / biotherapy) and has not been treated like this for at least 15 days

Inclusion criteria for population B: Henoch Schönlein purpura in remission

* The diagnosis of Henoch Schönlein purpura was made by a physician according to the EULAR / PRES / PRINTO 2010 criteria
* The patient has has a Henoch Schönlein purpura episode in the past, and no longer has any symptoms of the disease
* The patient is not treated via immunosuppression (steroids or other immunosuppressive / biotherapy) and has not been treated like this for at least 15 days

Inclusion criteria for population C: controls

* Subjects free from infectious, inflammatory or autoimmune diseases
* Candidates for elective surgery (circumcision, urological surgery, removal of tonsils and adenoids)

Exclusion Criteria:

* The patient is participating in another interventional study or is in an exclusion period determined by a previous study
* The child refuses to participate in the study
* Parents (or persons with parental responsibility if any) refuse to sign the consent
* It is impossible to correctly inform the patient or his/her parents (or persons with parental authority if any)
* The patient has another inflammatory or autoimmune disease
* Patient on immunosuppressive / biotherapy treatments

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Three different populations will be included in this study: (A) patients presenting with an acute episode of Henoch Schönlein purpura; (B) patients who have had an episode of Henoch Schönlein purpura in the past, but currently present with no symptoms; (C) a group of control patients recruted from elective surgery candidates at the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Percentage of blood Tregs | Day 0
Absolute Treg count | Day 0
  number / mm^3
Presence / absence of functional abnormality of plasma Tregs | Day 0

SECONDARY OUTCOMES:
Numerical abnormalities in other blood cell lines | Day 0
Serum cytokine levels | Day 0
  ng/ml
Serum IgA levels | Day 0
  mg/l
Presence/absence of bacterial translocation | Day 0
Quantification of bacterial translocation | Day 0
  (10^8 copies / µl)
Number of bacterial species detected in the intestinal microbiota | Day 0
Distribution of bacteria taxa present in the intestine among 3 categories | Day 0
  Bacteroidetes, Firmicutes and Actinobacteria

CONTACTS AND LOCATIONS:
Overall Officials: Tu Anh Tran, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Filleron A, Tran TA, Hubert A, Letierce A, Churlaud G, Kone-Paut I, Saadoun D, Cezar R, Corbeau P, Rosenzwajg M. Regulatory T cell/Th17 balance in the pathogenesis of paediatric Behcet disease. Rheumatology (Oxford). 2021 Dec 24;61(1):422-429. doi: 10.1093/rheumatology/keab253. PMID 33734346